CLINICAL TRIAL: NCT00946296
Title: Impact of SSKI Pre-Treatment on Blood Loss in Thyroidectomy for Graves Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11597
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-11

CONDITIONS: Graves Disease; Hyperthyroidism
Keywords: Graves Disease
MeSH Terms: conditions — Graves Disease; Hyperthyroidism | interventions — Potassium Iodide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Potassium Iodide (Active Comparator): 8 drops of Potassium Iodide in a glass of water, by mouth, daily for 7 days prior to operation.
  Interventions: Drug: Potassium Iodide
- No Treatment (No Intervention): The experimental group receives no treatment.

INTERVENTIONS:
Drug: Potassium Iodide — 8 drops of Potassium Iodide in a glass of water taken daily for 7 days prior to thyroidectomy. This is the current standard of care.
  Other Names: SSKI
  Arms: Potassium Iodide

SUMMARY:
The purpose of this study is to determine whether a brief course of SSKI (saturated solution of potassium iodide) administered preoperatively provides any benefit in the surgical management of patients undergoing thyroidectomy as definitive management of their Graves Disease.

DETAILED DESCRIPTION:
Historically Potassium Iodide was given to patients for 1 week prior to thyroidectomy. This common practice was used to decrease thyroid function and prevent thyroid storm during the thyroidectomy. However, in modern practice, nearly all patients presenting for surgical management have been made euthyroid through the use of medications such as propylthiouracil. Despite this potassium iodine continues to be administered with the presumption that it decreases the friability of the gland making surgery easier, with less blood loss.

The outcomes to be measured in this surgery are operative time, operative complications and blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a clinical diagnosis of Graves Disease
* Patients who have selected surgical resection as treatment of their Graves Disease
* Prior use of anti thyroid medication so that patient is clinically and biochemically euthyroid

Exclusion Criteria:

* Patients deemed unfit for surgery by operating surgeon or anesthesist
* Patients who are clinically hyperthyroid or have T3 or T4 levels 2X the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UMASS Memorial Health Care, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2005 and April 2013, subjects who had been determined to undergo thyroidectomy for definitive management of Graves Disease, were approached for participation in the study. Recruitment occurred in the endocrine practices of the investigators.
Period: Overall Study
Arm/Group | Potassium Iodide | No Treatment
Started | 21 | 15
Completed | 18 | 15
Not Completed | 3 | 0
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Potassium Iodide | No Treatment | Total
Number analyzed (Participants) | 21 | 15 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.44 (12.27) | 41.07 (10.62) | 40.25 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Blood Loss During Surgery
Description: Blood loss in milliliters during surgery.
Time Frame: up to 162 minutes
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Potassium Iodide | No Treatment
Number analyzed (Participants) | 18 | 15
mL | 61.67 (49.97) | 161.67 (134.62)

ADVERSE EVENTS:
Time Frame: 162 minutes
Description: During surgical procedure
Arm/Group | Potassium Iodide | No Treatment
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/15
Other Adverse Events (participants affected / at risk) | 0/21 | 0/15

LIMITATIONS AND CAVEATS:
Difficulty in enrolling subjects related to national shortages of potassium iodine which limited drug availability and contributed to delayed accrual as did decreased eligible patients and waning interest over time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No